CLINICAL TRIAL: NCT02128022
Title: Investigation Into Cardioprotective Effect of Glucagon-like Peptide-1 and it's Mechanism of Action During Myocardial Ischaemia
Brief Title: Cardioprotective Effects of GLP-1 and Their Mechanisms
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Papworth Hospital NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: P01900
Record Dates: First submitted 2014-04-24; First posted 2014-05-01 (Estimated); Last update posted 2016-04-11 (Estimated); Status verified 2016-04

CONDITIONS: Angina Pectoris
Keywords: Glucagon-Like Peptide 1; Angina Pectoris; Percutaneous Coronary Intervention; Ischemic Preconditioning; Myocardial Reperfusion Injury
MeSH Terms: conditions — Angina Pectoris; Myocardial Reperfusion Injury | interventions — glucagon-like peptide 1 (7-36)amide; Glyburide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- GLP-1 (7-36) amide and Glibenclamide (Experimental): Patients will receive 5mg Glibenclamide orally prior to PCI and infusion of GLP-1 (7-36) amide 1.2 pmol/Kg/min during PCI
  Interventions: Drug: GLP-1 (7-36) amide; Drug: Glibenclamide
- Glibenclamide alone (Experimental): Glibenclamide 5 mg orally prior to PCI
  Interventions: Drug: Glibenclamide
- GLP-1 (7-36) amide (Active Comparator): GLP-1 (7-36) amide
  Interventions: Drug: GLP-1 (7-36) amide
- Saline control (No Intervention): 0.9% saline only (no treatment with GLP-1 (7-36) amide or glibenclamide)

INTERVENTIONS:
Drug: GLP-1 (7-36) amide — Infusion of GLP-1 (7-36) amide 1.2 pmol/Kg/min
  Arms: GLP-1 (7-36) amide; GLP-1 (7-36) amide and Glibenclamide
Drug: Glibenclamide — Oral Glibenclamide 5mg
  Arms: GLP-1 (7-36) amide and Glibenclamide; Glibenclamide alone

SUMMARY:
Ischaemic heart disease is the most common cause of death in the UK. Glucagon-like peptide-1 (GLP-1) has been demonstrated to protect the heart when it is deprived of blood supply (ischaemia). The mechanism for this protection is not clear. Similar protection occurs with ischaemic conditioning of the heart, which is dependent on potassium channel opening.

The investigators intend to establish whether GLP-1 mediated protection shares a similar mechanistic pathway. In order to do this the investigators will measures pressure--volume loops generated in the main pumping chamber of the heart at the time of a percutaneous coronary intervention (stenting). Patients will be allocated to GLP-1 alone, GLP-1 with glibenclamide (a potassium channel blocking medication approved for human use), saline control or glibenclamide alone.

The investigators hypothesis is that the effect of GLP-1 will be abrogated by use of glibenclamide.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18
* Able to give informed consent
* Elective percutaneous intervention for a single vessel coronary stenosis
* Normal left ventricular function

Exclusion Criteria:

* Severe Co-morbidity
* Type 2 Diabetes Mellitus
* Nicorandil, Sulphonylureas, DPP4 inhibitors, GLP-1 agonists or Insulin use
* Women of child bearing age
* Myocardial infarction in previous three months
* Previous coronary artery bypass grafts

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2014-07; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Change in Isovlumetric Relaxation Constant - Tau (ms) | Measured at the time of procedure
  The isovolumetric relaxation constant, Tau, a measure of left ventricular diastolic function, will be measured during the second balloon occlusion of the coronary artery. This will be measured on pressure-volume loop using a conductance catheter.

SECONDARY OUTCOMES:
Left Ventricular Ejection Fraction (%) | Measured at the time of the procedure
  Ejection fraction, a measure of left ventricular systolic function, will be measured during the second balloon occlusion of the coronary artery. This will be measured on pressure-volume loop using a conductance catheter.
Maximal rate of change with time of left ventricular pressure - dP/dt max (mmHg/s) | Measured at the time of the procedure
  dP/dt max, a measure of left ventricular systolic function, will be measured during the second balloon occlusion of the coronary artery. This will be measured on pressure-volume loop using a conductance catheter.
Minimum rate of change with time of left ventricular pressure - dP/dt min (mmHg/s) | Measured at the time of procedure
  dP/dt min, a measure of left ventricular diastolic function, will be measured during the second balloon occlusion of the coronary artery. This will be measured on pressure-volume loop using a conductance catheter.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen P Hoole, MD, Principal Investigator — Papworth Hospital NHS Foundation Trust
Locations (1):
- Papworth Hospital, Cambridge, Cambridgeshire, United Kingdom

REFERENCES:
- [Derived] Giblett JP, Axell RG, White PA, Clarke SJ, McCormick L, Read PA, Reinhold J, Brown AJ, O'Sullivan M, West NE, Dutka DP, Hoole SP. Glucagon-like peptide-1 derived cardioprotection does not utilize a KATP-channel dependent pathway: mechanistic insights from human supply and demand ischemia studies. Cardiovasc Diabetol. 2016 Jul 19;15:99. doi: 10.1186/s12933-016-0416-3. PMID 27431258